CLINICAL TRIAL: NCT03941327
Title: Do AxoGuard Implants Decrease Shoulder Disability After Neck Dissections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-0212
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Spinal Accessory Nerve Injury; Cervical Lymphadenopathy
MeSH Terms: conditions — Accessory Nerve Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomly assigned to a control group or intervention group using a computer based randomization tool. Patient's undergoing bilateral neck dissection will receive an implant on one side and act as self control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Placebo Comparator): Patients who provide consent for implant placement but do not receive the implant.
  Interventions: Device: AxoGuard Nerve Cuff
- Interventional (Experimental): Patients who provide consent for implant placement and do receive the implant.
  Interventions: Device: AxoGuard Nerve Cuff

INTERVENTIONS:
Device: AxoGuard Nerve Cuff — A porcine collagen implant will be used to make a protective sheath around the participant's exposed spinal accessory nerve during surgery. This will be performed by physically wrapping the exposed nerve with the implant and suturing the ends together. The goal is to protect nerve from adhesions and compression in the absence of normal protective lymphatic soft tissue.

SUMMARY:
The purpose of this study is to determine whether Axoguard nerve protectors have a role in preventing shoulder disability and pain following spinal accessory nerve sparing neck dissections.

DETAILED DESCRIPTION:
The spinal accessory nerve is often manipulated during selective neck dissections in order to remove the fibrofatty tissues containing lymph nodes surrounding the nerve. Afterwards the nerve is left exposed without it's normal support making it vulnerable to adhesions, compression, and stretch injury. Axoguard nerve wraps have shown significant promise in preventing the recurrence of carpal tunnel following forearm surgery, and preventing impotence and incontinence following nerve sparing robotic radical prostatectomy. The investigators hypothesize that the same technology may aid in reducing shoulder disability and pain if used in spinal accessory nerve sparing neck dissections. In this prospective single blinded randomized controlled study the investigators will randomly assign patients to a control group that will not receive the AxoGuard nerve wrap, and a study group that will receive the AxoGuard nerve wrap around their exposed spinal accessory nerve(s) using a research randomization tool. The results will be stratified into groups including preoperative and postoperative stage of disease, preoperative and postoperative nodal (neck) stage, history of radiation, and whether or not level 2B was dissected. Individuals with a history of pre-existing disabling shoulder complaints, individuals under the age of 18, individuals who cannot provide their own informed consent, and individuals undergoing a neck dissection that will remove the sternocleidomastoid muscle or spinal accessory nerve will be excluded from the study. Patients will undergo preoperative shoulder assessment using the Constant-Murley shoulder outcome score at their initial clinical visit. Postoperative outcomes will be recorded at 2 weeks, 2 months, 4 months, and 6 months and measured by the Shoulder Disability Questionnaire, Rand-36 quality of life survey, pain scale, and Constant-Murley shoulder outcome score. With this study the investigators aim to show a clinically significant improvement in shoulder function following spinal accessory nerve sparing neck dissections when AxoGuard nerve wraps are used to protect the nerve. Additionally, the investigators aim to improve patient satisfaction, decrease post-op pain, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

-Any neck dissection (cervical lymphadenectomy) that involves resection of level 2 cervical lymph nodes for malignancy and does not fall into the categories listed under the exclusion criteria.

Exclusion Criteria:

1. History of modified radical neck dissection involving removal of spinal accessory nerve or sternocleidomastoid muscle
2. History of radical neck dissection
3. History of pre- existing disabling shoulder complaints
4. <18 years of age
5. Any individual unable to provide consent for his/her self.
6. Any individual with allergy, sensitivity, or aversion to porcine material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder function | The comparison of improvement or change in shoulder function over 6 months between the control and intervention groups will be the primary outcome measure.
  Shoulder function will be assessed by Constant-Murley shoulder scale. The Constant-Murley shoulder scale is a validated subjective and objective survey of overall shoulder function. The scale ranges from 0 (no shoulder function) to 100 (perfect shoulder function). It consists of several questions about pain and disability as well as actual shoulder testing that will be performed by the consenting physician during the participant's clinic appointment.

SECONDARY OUTCOMES:
Postoperative pain following neck dissection: rate shoulder pain from 1-10 | Patients will be asked to rate shoulder pain from 1-10 at each postoperative visit over the course of 6 months.
  The comparison of the improvement or change in pain scores over 6 months between the control group and intervention group will be assessed at each clinical visit over the course of 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided